CLINICAL TRIAL: NCT02064205
Title: A Double Blind, Placebo Controlled, Randomized, Cross-over Study to Assess the Effects of Polydextrose on Appetite Suppression and Its Mechanisms of Action in Healthy Women With a Normal Weight and Overweight Female Participants.
Brief Title: Appetite Suppression Trial With Polydextrose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: W.J. Pasman (Other)
Responsible Party: Sponsor-Investigator, W.J. Pasman, Project Manager Clinical Trials, TNO
Organization: TNO (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: JZ PDX Satiety; WM-01-2014 (Other: QPS, The Netherlands)
Record Dates: First submitted 2014-02-11; First posted 2014-02-17 (Estimated); Results first posted 2016-07-27 (Estimated); Last update posted 2022-06-06 (Actual); Status verified 2022-05

CONDITIONS: Body Weight; Non-restrained Eaters
Keywords: pre-load; satiety; energy intake; appetite
MeSH Terms: conditions — Body Weight | interventions — polydextrose; High Fructose Corn Syrup

STUDY DESIGN:
Intervention Model Description: Breakfast meal with or without polydextrose
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- polydextrose or glucose syrup at breakfast (Active Comparator): Breakfast with pre-load four hours before lunch
  Interventions: Dietary Supplement: 12.5 g polydextrose; Dietary Supplement: glucose syrup
- Pre-load with yogurt and polydextrose or glucose later (Placebo Comparator): Breakfast without pre-load. Pre-load with yogurt provided 1.5h before lunch.
  Interventions: Dietary Supplement: 12.5 g polydextrose; Dietary Supplement: glucose syrup

INTERVENTIONS:
Dietary Supplement: 12.5 g polydextrose — Appetite suppressing supplement is added in yogurt and provided with breakfast (four hours before lunch) or 1.5h before lunch. Also yogurt with control (glucose syrup) is tested for its satiating effect.
  Other Names: Litesse®Ultra TM
Dietary Supplement: glucose syrup — Glucose syrup is used a control product for the polydextrose

SUMMARY:
Overweight and obesity are a global epidemic, which causes a rapid increase in the frequency of diabetes and cardiovascular diseases. Food ingredients that influence the mechanisms that regulate satiety may play a role in weight management. Suppression of appetite may reduce energy intake, which in return may lead to body weight reduction. This study aims to verify the appetite suppressive effect of polydextrose in comparison to a placebo in normal weight and overweight women.

DETAILED DESCRIPTION:
Polydextrose is a well-tolerated, low calorie glucose polymer (4kJ/g) that can be easily incorporated into various food applications to replace sugar and fat (Auerbach et al., 2007). Polydextrose is poorly digested in the upper gastrointestinal tract and therefore shows fiber-like properties. The addition of polydextrose to foods may increase the satiating properties of foods.

Previous studies have shown that:

* Consuming polydextrose-containing preloads (6.25 - 25.0 g polydextrose) resulted in a significant lower energy intake at lunch compared to the control (Astbury et al., 2013; Ranawana et al., 2013; Hull et al., 2012; King et al., 2005).
* Polydextrose is able to modify appetite ratings at low (6.25 - 12.5 g polydextrose) (Hull et al., 2012) and high doses (56.7 g/d) (Konings et al., 2013).
* Polydextrose (15.0 g) induced enhanced GLP-1 response after a high-fat meal in obese participants (Tiihonen et al., 2012).

Therefore, it is hypothesized that with the consumption of 12.5 g polydextrose as compared with the placebo, appetite will be suppressed, resulting in:

* a lower consumption at lunch (energy intake at lunch)
* change in appetite scores (VAS)
* change in satiety hormones (CCK, PYY, GLP-1, ghrelin)
* change in glucose and insulin
* change in stomach emptying rate
* change in gastric wellbeing

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, female participants aged 20-45 years inclusive
2. BMI: 20-30 kg/m2 inclusive
3. Written consent regarding participation after full information regarding all details of the study
4. Normal Dutch eating habits (consuming mostly three main meals per day; used to eat bread for lunch)

Exclusion Criteria:

1. Pregnancy
2. On-going or recent treatment for diabetes, hypertension, coronary heart disease, psychiatric conditions, inflammatory chronic disease - rheumatoid arthritis, Crohn Disease, ulcerous colitis, chronic constipation, eating disorders, or any disease condition which interferes with ADME of the investigational product
3. Reported postmenopausal
4. Having menstruation problems, e.g. PCOS
5. Reported to be on a slimming diet or other dietary treatment (currently or during last two months, like vegetarian diet, lactose restricted diet etc.)
6. Aversion towards products (yoghurt) provided in the study
7. On-going use of any slimming preparations
8. Any kind of dysfunction of digestive tract, food allergy, chronic constipation, recent/actual gastroenteritis
9. Restrained eaters (score DEBQ >3.4)
10. Participants consuming more than 23g of dietary fiber per day - P75 according to the Dutch National Food Consumption Survey - (as assessed with a general short questionnaire which gives estimation on the fiber intake. Exact fiber intake will not be calculated)
11. Smoker in the last 3 months
12. Heavy coffee drinkers (more than 6 cups a day)
13. High level of physical activity: Participants who perform more than 3 hours of intense training/sport activity per week (this will not include normal cycling transport)
14. Heavy alcohol consumers, no more than 14 units per week (1 unit represents 1 standard glass/portion of alcohol, independent of the type of alcoholic drink).

Remark:

When enough subjects are eligible (> 32), the women with the highest BMI will be selected to participate. At least 50% of the subjects will have a BMI ranging of 25-30. Also at least 50% of the women will be in the age range of 25-45 years. When more than 32 subjects are eligible the eldest subjects will be included.

With respect to eligibility of the subjects:

the BMI criterion always comes for age criterion, meaning that overweight is stressed to be of more importance for this study than age. Overweight will always come first, even when already > 50% of the women with a BMI 25-30 have been included. In this way the overweight group of women will be studied as much as possible.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2014-05; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naguib Muhsen, MD, Principal Investigator — QPS, The Netherlands
Locations (1):
- QPS, Groningen, Netherlands

REFERENCES:
- [Derived] Ibarra A, Olli K, Pasman W, Hendriks H, Alhoniemi E, Raza GS, Herzig KH, Tiihonen K. Effects of polydextrose with breakfast or with a midmorning preload on food intake and other appetite-related parameters in healthy normal-weight and overweight females: An acute, randomized, double-blind, placebo-controlled, and crossover study. Appetite. 2017 Mar 1;110:15-24. doi: 10.1016/j.appet.2016.12.002. Epub 2016 Dec 2. PMID 27916475

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment lasted from May 2014 - August 2014. 121 subjects were planned for screening. 46 subjects met the inclusion criteria, 37 subjects did not show up, and 38 subjects had screening failures.
  The CRO that conducted the clinical trial was:
  QPS Netherlands B.V. Groningen The Netherlands
Pre-assignment Details: In the study four test days were conducted, one weekly. Between test day there are six days of wash-out.
Groups:
- All Study Participants: A: Breakfast with the pre-load and 12.5 g polydextrose B:Breakfast with the pre-load without polydextrose C: Breakfast and pre-load with 12.5 g polydextrose at 150 min D:Breakfast and pre-load without polydextrose at t=150 min
  Eight orders:
  A-B-D-C; B-C-A-D; C-D-B-A; D-A-C-B; A-D-B-C; C-B-D-A; B-A-C-D; D-C-A-B.
Period: Overall Study
Arm/Group | All Study Participants
Started | 32
Condition A | 32
Condition B | 32
Condition C | 31
Condition D | 32
Completed | 31
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Overall Baseline Charactistics of 32 Slightly Overweight Women: Baseline data of the subjects were measured at screening at least one week before the start of the study.
Arm/Group | Overall Baseline Charactistics of 32 Slightly Overweight Women
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.4 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 0
Region of Enrollment [Number; unit: participants]
  Netherlands | 32
Body weight [Mean (Standard Deviation); unit: kg] | 74.4 (7.8)
Height [Mean (Standard Deviation); unit: meter] | 1.70 (0.04)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index
  kg/m^2 | 25.9 (2.7)
BPsys [Mean (Standard Deviation); unit: mm Hg] — Systolic blood pressure
  mm Hg | 113.5 (9.9)
BPdia [Mean (Standard Deviation); unit: mm Hg] — Diastolic blood pressure
  mm Hg | 64.2 (9.0)
Dutch Eating Restraintness Score [Mean (Standard Deviation); unit: units on a scale] — Score ranges from 0 - 5 0 = unrestrained 5 = very restrained
  units on a scale | 2.4 (0.4)
Dietary fiber intake [Mean (Standard Deviation); unit: grams/day] | 18 (4)

OUTCOME MEASURES:

1. Primary Outcome: Energy Intake at an ad Libitum Lunch on a Test-day in Normal Weight and Overweight Women.
Description: Yogurt with a polydextrose (fiber with satiating effect) is consumed in the morning with breakfast or later in the morning. The satiating effect of the addition of polydextrose is tested on the amount of food consumed with lunch four hours or 1.5h later.
Time Frame: Four hours or 1.5 hour after consumption of a pre-load at up to day 22
Population: Energy intake
Measure: Mean (Standard Deviation); unit: kJ
Groups:
- Polydextrose Syrup at Breakfast [A]: Breakfast with pre-load four hours before lunch
  12.5 g polydextrose: Appetite suppressing supplement is added in yogurt and provided with breakfast, four hours before lunch.
- Glucose Syrup at Breakfast (Control) [B]: Breakfast with control pre-load four hours before lunch
  Yogurt with control (glucose syrup) is tested for its satiating effect.
  glucose syrup: Glucose syrup is used a control product for the polydextrose
- Pre-load With Polydextroseglucose Before Lunch [C]: Breakfast without pre-load. Pre-load with yogurt and polydextrose provided 1.5h before lunch.
  12.5 g polydextrose: Appetite suppressing supplement is added in yogurt 1.5h before lunch.
- Pre-load With Yogurt and Glucose Before Lunch [D]: Breakfast without pre-load. Pre-load with yogurt and glucose (control) provided 1.5h before lunch.
  Yogurt with control (glucose syrup) is tested for its satiating effect 1.5h before lunch
Arm/Group | Polydextrose Syrup at Breakfast [A] | Glucose Syrup at Breakfast (Control) [B] | Pre-load With Polydextroseglucose Before Lunch [C] | Pre-load With Yogurt and Glucose Before Lunch [D]
Number analyzed (Participants) | 31 | 31 | 31 | 31
kJ | 2694 (1028) | 2537 (933) | 2317 (940) | 2335 (1051)
Statistical Analysis 1: Comparison: Pre-load With Polydextroseglucose Before Lunch [C] vs Pre-load With Yogurt and Glucose Before Lunch [D]; A mixed model was applied to analyze the Energy Intakes (ad libitum lunch and daily) were done one-sided to evaluate the appetite suppressive effect after the pre-load snack (condition C versus D); Test type: Superiority or Other; p = 0.2918, Mixed Models Analysis; Mean Difference (Final Values) = 18, Standard Deviation 1000

2. Secondary Outcome: The Appetite Suppressive Effect of Polydextrose During Meal Consumption (Satiation) and Satiety (After Food Consumption)
Description: The appetite suppressive effect of polydextrose measured with Visual Analogue rating Scales (VAS). The AUCs were calculated for the scores obtained before - first score after meal intake (satiation) and for score after meal till start of next meal (in between meals, satiety). The VAS scores ranged from 0-100 for hunger and fullness (HUNGER: 0 = no hunger , 100 = very hungry; FULNESS: 0 = not full, 100 = very full)
Time Frame: one day
Measure: Mean (Standard Deviation); unit: mm*min
Groups:
- Polydextrose Syrup Preload With Yogurt With Breakfast [A]: Polydextrose syrup preload with yogurt with breakfast was consumed four hours before lunch
- Glucose Syrup as Proload With Breakfast (Control) [B]: Breakfast with glucose syrup and yogurt provided four hours before lunch.
- Pre-load With Polydextrose Before Lunch [C]: Pre-load with polydextrose syrup and yogurt is provided 1.5h before lunch
- Pre-load With Glucose Syrup Before Lunch [D]: Pre-load with glucose syrup and yogurt was provided 1.5h before lunch.
Arm/Group | Polydextrose Syrup Preload With Yogurt With Breakfast [A] | Glucose Syrup as Proload With Breakfast (Control) [B] | Pre-load With Polydextrose Before Lunch [C] | Pre-load With Glucose Syrup Before Lunch [D]
Number analyzed (Participants) | 32 | 32 | 31 | 31
mm*min
  Hunger score | 358.3 (183.4) | 336.8 (158.9) | 356.7 (169.1) | 280.2 (167.2)
  Fullness score during first phase | -424.7 (192.4) | -443.0 (190.7) | -326.6 (207.6) | -308.2 (155.6)
  Hunger score (satiety period) | 4898.9 (3424) | 4134.9 (2962.9) | 962.8 (1232.2) | 592.9 (987.2)
  Fulness score (satiety period) | -6009.9 (3670.8) | -5048.3 (4088.4) | -734.8 (1263.5) | -1077.4 (1118.1)
Statistical Analysis 1: Comparison: Pre-load With Polydextrose Before Lunch [C] vs Pre-load With Glucose Syrup Before Lunch [D]; AUC of hunger scores before preload intake for condition C versus D; Test type: Superiority or Other; p = 0.0109, Mixed Models Analysis

3. Secondary Outcome: Evaluate Effect of Pre-load on Satiety Hormones in Normal Weight and Overweight Women.
Description: The satiety hormones CCK, GLP-1, ghrelin and PYY are measured before (t=0) and after breakfast consumption (at t=30, 60, 90, 150, 240) . This is done on day 01, day 08, day 15 and day 22 with at least four days wash-out in-between.
  The satiety hormones were only measured in the conditions when the pre-load was given with breakfast (condition A and B).
  Area under the curves were calculated of the time curves.
Time Frame: Four hour curves (t=0, 30, 60, 90, 150 and 240 min) of day 01, day 08, day 15 and day 22.
Population: Only in condition A and B blood was drawn and satiety hormones were analyzed.
Measure: Mean (Standard Deviation); unit: (mcg*min)/mL
Groups:
- Polydextrose Syrup at Breakfast [A]: Breakfast with polydextrose and yogurt provided four hours before lunch.
- Glucose Syrup at Breakfast (Control) [B]: Breakfast with glucose syrup and yogurt provided four hours before lunch.
Arm/Group | Polydextrose Syrup at Breakfast [A] | Glucose Syrup at Breakfast (Control) [B]
Number analyzed (Participants) | 32 | 32
(mcg*min)/mL
  CCK (AUC) | 241.15 (113.69) | 265.03 (112.44)
  Ghrelin (AUC) | -23479 (33428) | -20902 (21150)
  PYY (AUC) | 1745.5 (2861.7) | 1210.5 (2832.6)
  GLP-1 (AUC) | 447.65 (298.11) | 316.02 (244.98)
Statistical Analysis 1: Comparison: Polydextrose Syrup at Breakfast [A] vs Glucose Syrup at Breakfast (Control) [B]; A mixed model was applied to statistically analyze satiety hormones having Conditions and Time as a fixed factor and having Subject, Cohort, and Treatment Day as random factors; Test type: Superiority or Other; p = 0.0216, Mixed Models Analysis — GLP-1

ADVERSE EVENTS:
Time Frame: During the conduct of the study; June - November 2014
Groups:
- Condition A: Breakfast with preload of yogurt and polydextrose
- Condition B: Breakfast with preload of yogurt and glucose control
- Condition C: Breakfast without preload; pre-load provided at t=150 min as a mid-morning snack of yogurt and polydextrose
- Condition D: Breakfast without preload; pre-load provided at t=150 min as a mid-morning snack of yogurt and glucose syrup
Arm/Group | Condition A | Condition B | Condition C | Condition D
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32 | 0/31 | 0/32
Other Adverse Events (participants affected / at risk) | 5/32 | 5/32 | 2/31 | 2/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Condition A (N=32) | Condition B (N=32) | Condition C (N=31) | Condition D (N=32)
Headache (Nervous system disorders) | 2 | 0 | 2 | 1
Nausea (Gastrointestinal disorders) | 2 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomitting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Presyncope (light headedness) (Nervous system disorders) | 1 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0
catheter site pain (General disorders) | 0 | 1 | 0 | 0
Pyrexia (fever) (General disorders) | 0 | 1 | 0 | 0
Infections and infestations (Infections and infestations) | 0 | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Dysmenorrhea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No